CLINICAL TRIAL: NCT04450082
Title: One Anastomosis Gastric Bypass After Sleeve Gastrectomy Failure: Does a Single Procedure Fit for All?
Brief Title: One Anastomosis Gastric Bypass After Sleeve Gastrectomy Failure
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, Head of Bariatric Unit, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 22062020; 22062020 (Other: Redosurgery)
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Bariatric Surgery Candidate
Keywords: Sleeve gastrectomy; One Anastomosis gastric bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- One anastomosis gastric bypass: One anastomosis gastric bypass in Sleeve Gastrectomy failure
  Interventions: Procedure: One anastomosis gastric bypass

INTERVENTIONS:
Procedure: One anastomosis gastric bypass — The linear stapler divides the stomach horizontally at the junction of the corpus and antrum at the level of crow's foot. In cases where the pre-operative study has shown the presence of the gastric fundus, if possible the fundus was dissected and a long, narrow gastric pouch was designed starting from beyond the crow's foot to just lateral the angle of His over a 42-Fr orogastric tube. Gastrojejunostomy was then performed between 200-220 cm distally to the ligament of Treitz using a 45-mm.

SUMMARY:
This study is a retrospective analysis of prospectively collected data on 582 obese patients. The primary aim of the study was to evaluate %Excess Weight Loss, Body Mass Index (BMI) and remission of comorbidity at mid- and long-term follow-up after One Anastomosis Gastric Bypass in subjects previously underwent Sleeve Gastrectomy. The secondary aim was to investigate the onset of esophagitis and gastritis at Upper Endoscopy (UE) and the presence of nutritional deficiencies in patients undergoing One Anastomosis Gastric Bypass as a redo surgery

DETAILED DESCRIPTION:
This study is a retrospective analysis of prospectively collected data on 582 obese patients. It was conducted according to the ethical principles stated in the Declaration of Helsinki. Written informed consent was obtained from all subjects. The study protocol was approved by the Regional Ethics Committee. From January 2014 to February 2019, morbid obesity patients who failed previous treatment with SG and referred to our bariatric center in the Department of General and Emergency Surgery of "A. Rizzoli" Hospital in Lacco Ameno (Naples, Italy) for a new bariatric procedure, were considered in the study. Redo surgery was only considered if patients still met the criteria for primary bariatric surgery according to guidelines [body mass index (BMI) >35 kg/m2 with co-morbidities, BMI >40 kg/m2] at the time clinical and anthropometrical revision8. A postoperative follow-up of at least 24 months was also considered inclusion criteria. Exclusion criteria were as follows: patients in whom Sleeve Gastrectomy was already performed as revision surgery; patients underwent any other abdominal surgical procedure after One Anastomosis Gastric Bypass not correlated to the bariatric procedure, the presence at baseline of esophagitis B according to the Los Angeles scale, Hiatal Hernia (HH) > 5 cm and history of GERD-related symptoms (i.e., heartburn, pyrosis, regurgitation) not responsive to proton pump inhibitors and/or severe Lower Esophageal Sfinter incontinence. All procedures were performed by the same experienced bariatric surgeons.

Pre-operative evaluation All patients underwent a multidisciplinary preoperative evaluation including anthropometric measurements (height in cm, weight in kg, Body Mass Index in kg/m2), comorbidity evaluation, preoperative Upper Endoscopy with Helicobacter Pylori test, abdomen ultrasound, chest x-ray and nutritional status evaluation.

Radiographic barium swallow test was performed for the diagnosis of HH or presence of gastric fundus. Barium swallow X-ray protocol consisted of five swallows of barium always using the same amount of liquid; anteroposterior and oblique views were obtained in upright and supine positions. Measurements were done using a standardized protocol: a distance of more than 2 cm between the gastroesophageal junction and the diaphragmatic hiatus was defined as a sliding Hiatal Hernia. Preoperative assessments of patient eligibility for bariatric surgery included consultation with the multidisciplinary committee (surgeon, radiologist, diabetologist and psychiatrist) to exclude patients with non-adjusted eating patterns or eating disorders.

Failure of Sleeve Gastrectomy was defined as a consequence of Insufficient Weight Loss or Weight Regain. Insufficient Weight Loss or Weight Regain were analyzed considering the modifications of the percentage of excess weight loss <50% and/or the percentage of total weight loss <25%. A failure of Sleeve Gastrectomy was recognized if the subject was not able to reduce the Body Mass Index <35 with the persistence of co-morbidity or Body Mass Index <40 at least 2-year after the primary surgery.

ELIGIBILITY:
Inclusion criteria:

* informed consent.
* morbid obesity defined as body mass index (BMI) 40 kg/m2
* Sleeve Gastrectomy failure

Exclusion Criteria:

* previous bariatric surgical procedures other than Sleeve Gastrectomy
* endocrine disorders causing obesity
* pregnancy or lactation
* psychiatric illness
* inflammatory bowel disease
* Barrett ́s oesophagus
* severe gastro-oesophageal Reflux Disease with esophagitis B and C
* a large hiatal hernia (>5 cm)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent to One anastomosis gastric bypass after sleeve gastrectomy failure
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2020-06-21 (Actual)

PRIMARY OUTCOMES:
Body Mass Index (kg/m2) | 24 months
  Body Mass Index (kg/m2) at follow-up after OAGB in subjects previously underwent Sleeve Gastrectomy

SECONDARY OUTCOMES:
Gastroesophageal reflux disease(GERD) | at 24 months
  Esophagitis grading according to Los Angeles classification with Upper endoscopy (Grade A: One or more mucosal breaks < 5 mm in maximal length; Grade B: One or more mucosal breaks > 5mm, but without continuity across mucosal folds; Grade C: Mucosal breaks continuous between ≥ 2 mucosal folds, but involving less than 75% of the esophageal circumference Grade D Mucosal breaks involving more than 75% of esophageal circumference

IPD SHARING:
Plan to Share IPD: No